CLINICAL TRIAL: NCT03050372
Title: Double-Blind, Sham-Controlled Crossover Pilot Study of Low Field Magnetic Stimulation (LFMS) on Subjective and Objective Measures of Sleep
Brief Title: Study of Low Field Magnetic Stimulation (LFMS) on Measures of Sleep
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding no longer available
Sponsor: Medical University of South Carolina (Other)
Collaborators: Tal Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00055979
Record Dates: First submitted 2016-12-16; First posted 2017-02-10 (Actual); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Insomnia, Primary
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Low Field Magnetic Stimulation (Experimental): LFMS - Active
  Interventions: Device: LFMS - Active
- Sham Low Field Magnetic Stimulation (Sham Comparator): LFMS - Sham
  Interventions: Device: LFMS - Sham

INTERVENTIONS:
Device: LFMS - Active — A non-invasive form of brain stimulation administered from a device resembling a bird cage. The device covers the top part of the head for the duration of stimulation (in the current study, 20 minutes)
  Arms: Active Low Field Magnetic Stimulation
Device: LFMS - Sham — A simulation of the LFMS-Active intervention, using the same device that produces a sound similar to the sound made by the device during the active treatment, for a similar duration (in the current study, 20 minutes)
  Arms: Sham Low Field Magnetic Stimulation

SUMMARY:
Participants will be recruited and screened through ongoing studies in the sleep and anxiety disorders clinic. Participants with insomnia will be consented to complete several questionnaires, undergo a brief physical exam, provide a urinalysis, and undergo 5 nights of active or sham Low Field Magnetic Stimulation (LFMS) followed by an overnight sleep study. Each of the two treatment conditions (active versus sham) will be conducted on two consecutive nights. There will be no more than 7 days between the adaptation night and the first treatment condition and no more than 7 nights between each of the two-night treatment conditions . Thus, each participant who completes the full study will spend a total of 5 nights in the sleep laboratory and the time interval from the first adaptation night to completion of the study may range from 5-19 days for any particular individual.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia diagnosis per DSM-5 criteria
* Performing tasks in a timely manner (compared to the person's usual level of performance)
* Pittsburgh Sleep Quality Index (PSQI) > 6 and one of the following:
* Sleep Efficiency < 85% (per Consensus Sleep Diary)
* Insomnia Severity Index (ISI) score > 15
* Sleep latency (subjective) and/or time awake after sleep onset (subjective) >30 minutes.
* Not currently depressed (previous major depressive episodes and current antidepressant medication permitted as long as remission and current medication dosage has been stable for ≥ 1 month).
* Willing to refrain from alcohol for twenty-four hours before presenting to sleep lab for sleep studies
* BMI > 18 and < 50 kg/m2

Exclusion Criteria:

* Current major depressive episode
* Current substance-induced depressive disorder
* Self-reported use of benzodiazepines or hypnotic drugs in last two weeks
* Self-reported use of marijuana in previous 72 hours
* Alcohol Use Disorders Identification Test (AUDIT) score > 10
* Fagerstrom Test for Nicotine Dependence (FTND) score > 4
* Insomnia limited to early morning awakening (without difficulty initiating or maintaining sleep),
* Narcolepsy
* Seizure Disorder (not including childhood febrile seizures)
* Recent treatment with anticonvulsant medications
* Obstructive or central sleep apnea
* Circadian rhythm sleep-wake disorders
* Recurrent isolated sleep paralysis
* Current substance-induced insomnia
* Chronic pain disorder
* Daily Caffeine Consumption > 500 mg/d (Uhde, 1989)
* Restless legs syndrome
* Periodic Leg Movement Disorder
* Benzodiazepines or antipsychotic medications during past 30 days
* Presence of drugs of abuse (excluding marijuana, urinalysis)
* Pregnancy or plans to become pregnant
* History of severe allergic reactions to adhesive tape
* History of neurological disorder
* Conductive, ferromagnetic or other magnetic-sensitive metals in the head, neck, chest, upper arms, or any area that will be within 18 inches of the treatment coil.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Uhde, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
This process is still being discussed by investigators. Once plan is complete it will likely include protocol and primary outcome measures which may be accessed through peer reviewed publications.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility screening was completed over the phone by trained sleep personnel; sleep laboratory is located at the Medical University of South Carolina's Institute of Psychiatry at 67 President St., Charleston S.C. This is a crossover study; each participant is exposed to both active and sham conditions.
Pre-assignment Details: N=209 subjects screened from 07/2016-07/2017; N=193 participants were excluded prior to PSG because they declined to participate (N=49), did not meet the age criterion (N=28), did not meet the sleep criterion (N=61), had co-morbid psychiatric disorders (N=42), or for other reasons (N=13); N=4 excluded after consent due to medication/baby/no-show.
Groups:
- Active Low Field Magnetic Stimulation (LFMS), Then Sham LFMS: Adaptation Night; then two consecutive nights of Active LFMS; after washout two consecutive nights of Sham LFMS
  LFMS - Active: A non-invasive form of brain stimulation administered from a device resembling a bird cage. The device covers the top part of the head for the duration of stimulation (in the current study, 20 minutes); then participants complete a full night of sleep in the sleep lab
  LFMS - Sham: A simulation of the LFMS-Active intervention, using the same device that produces a sound similar to the sound made by the device during the active treatment, for a similar duration (in the current study, 20 minutes); then participants complete a full night of sleep in the sleep lab
- Sham Low Field Magnetic Stimulation (LFMS), Then Active LFMS: Adaptation Night; then two consecutive nights of Sham LFMS; after washout followed by two consecutive nights of Active LFMS
  LFMS - Active: A non-invasive form of brain stimulation administered from a device resembling a bird cage. The device covers the top part of the head for the duration of stimulation (in the current study, 20 minutes); then participants complete a full night of sleep in the sleep lab
  LFMS - Sham: A simulation of the LFMS-Active intervention, using the same device that produces a sound similar to the sound made by the device during the active treatment, for a similar duration (in the current study, 20 minutes); then participants complete a full night of sleep in the sleep lab
Period: Adaptation Night (Night #1 PSG)
Arm/Group | Active Low Field Magnetic Stimulation (LFMS), Then Sham LFMS | Sham Low Field Magnetic Stimulation (LFMS), Then Active LFMS
Started | 6 | 6
Completed | 5 (N=1 subject removed from study due to mild sleep apnea during adaptation night) | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: First Intervention (Nights #2 and #3)
Arm/Group | Active Low Field Magnetic Stimulation (LFMS), Then Sham LFMS | Sham Low Field Magnetic Stimulation (LFMS), Then Active LFMS
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Second Intervention (Nights #4 and #5)
Arm/Group | Active Low Field Magnetic Stimulation (LFMS), Then Sham LFMS | Sham Low Field Magnetic Stimulation (LFMS), Then Active LFMS
Started | 5 | 6
Completed | 5 | 5 (N=1 subject (blind only broken after double-blind analysis) moved out off State; lost to study)
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants are randomized to receive either two consecutive nights of "Active Low Field Magnetic Stimulation" followed by "Sham Low Field Magnetic Stimulation" or vice versa.
  Active Low Field Magnetic Stimulation LFMS - Active: A non-invasive form of brain stimulation administered from a device resembling a bird cage. The device covers the top part of the head for the duration of stimulation (in the current study, 20 minutes)
  Sham Low Field Magnetic Stimulation LFMS - Sham: A simulation of the LFMS-Active intervention, using the same device that produces a sound similar to the sound made by the device during the active treatment, for a similar duration (in the current study, 20 minutes)
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.58 (8.512)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Height [Mean (Standard Deviation); unit: inch] | 67.83 (3.54)
Weight [Mean (Standard Deviation); unit: lbm (pound mass)] | 184.83 (35.70)
PSQI (Pittsburgh Sleep Quality Inventory) [Mean (Standard Deviation); unit: units on a scale] — Pittsburgh Sleep Quality Inventory (PSQI) is a well established 10-question questionnaire (24 items incl. sub-questions 5a-j and 10a-e) that assesses subjective sleep quality, -latency, -duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, daytime dysfunction. Individual items' responses are in the range of 0-3; a total PSQI score is derived by first deriving 7 equally weighted components from all 24 responses; each component is in the range of 0-3, resulting in a total score (sum of all components) of 0-21; a total PSQI score of >=5 is associated with poor sleep.
  units on a scale | 11.58 (2.68)

OUTCOME MEASURES:

1. Primary Outcome: Sleep Onset Latency (SOL) After Sham vs. Active LFMS (Each Averages of Two Consecutive Nights); and Difference From Baseline (Adaptation Night)
Description: SOL is the time of transition from wake to sleep (non-REM S1) measured in minutes; a validated objective measure extracted directly from full-night polysomnography (PSG). SOL of 0-5min is associated with severe sleep deprivation; 5-10min is moderate sleep debt; 10-15min indicates mild sleep debt; 15-20min is little-to-no sleep debt; and >20min is considered to be associated with no sleep debt.
Time Frame: Each night (5 nights total): Baseline (adaptation night #1), First Intervention (nights #2,#3), Second Intervention (nights #4,#5); Interventions randomized Sham or Active LFMS
Population: 12 subjects completed the adaptation night (Baseline); 1 subject was then excluded due to mild sleep apnea; 11 subjects completed treatment (active or sham) nights 1/2; 1 subject moved out of State (received sham in night 1/2); 10 subjects completed all 5 nights: adaptation night and intervention nights 2/3 & 4/5, each pair either sham or active.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
minutes
  Baseline SOL | 43.35 (25.95) | 43.35 (25.95)
  Intervention LFMS; two-night average in each arm | 53.88 (40.03) | 46.35 (34.50)
  Change from Baseline SOL | 10.53 (31.67) | 3.00 (22.77)
Statistical Analysis 1: Comparison: Active Low Field Magnetic Stimulation vs Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of SOL for active/sham LFMS are equal; Ha: Means differ Note this paired t-test is equivalent to: H0: Mean changes from Baseline SOL for active/sham LFMS are equal Ha: Means differ; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.329, t-test, 2 sided
Statistical Analysis 2: Comparison: Active Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of SOL for Baseline and Active LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline SOL for Active LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.321, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of SOL for Baseline and Sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline SOL for Sham LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.687, t-test, 2 sided

2. Primary Outcome: Wake After Sleep Onset (WASO) After Sham vs. Active LFMS (Each Averages of Two Consecutive Nights); and Difference From Baseline (Adaptation Night)
Description: Total time awake after initial sleep onset in minutes; validated objective measure directly extracted from polysomnography (PSG); we average measures from both consecutive nights under each of the two interventions (Sham or Active LFMS)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
minutes
  Baseline WASO | 80.85 (78.41) | 80.85 (78.41)
  Sham or Active LFMS (two-night average) | 54.80 (46.87) | 56.00 (31.31)
  Change from Baseline WASO | 26.05 (41.69) | 24.85 (59.75)
Statistical Analysis 1: Comparison: Active Low Field Magnetic Stimulation vs Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of WASO for active/sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to: H0: Mean changes from Baseline WASO for active/sham LFMS are equal Ha: Means differ; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.925, t-test, 2 sided
Statistical Analysis 2: Comparison: Active Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of WASO for Baseline and Active LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline WASO for Active LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.08, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of WASO for Baseline and Sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline WASO for Sham LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.221, t-test, 2 sided

3. Primary Outcome: Total Sleep Time (TST) After Sham vs. Active LFMS (Each Averages of Two Consecutive Nights); and Difference From Baseline (Adaptation Night)
Description: Total Sleep Time is the total time spent sleeping (non-wake stages S1-S5) in minutes; validated objective measure directly extracted from polysomnography (PSG).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
minutes
  Baseline TST | 359.60 (86.60) | 359.60 (86.60)
  Sham or Active LFMS (two-night average) | 370.40 (80.96) | 388.53 (73.02)
  Change from Baseline TST | 10.80 (60.50) | 28.93 (82.73)
Statistical Analysis 1: Comparison: Active Low Field Magnetic Stimulation vs Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of TST for active/sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to: H0: Mean changes from Baseline TST for active/sham LFMS are equal Ha: Means differ; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.197, t-test, 2 sided
Statistical Analysis 2: Comparison: Active Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of TST for Baseline and Active LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline TST for Active LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.586, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of TST for Baseline and Sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline TST for Sham LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.298, t-test, 2 sided

4. Primary Outcome: Sleep Efficiency (SE) After Sham vs. Active LFMS (Each Averages of Two Consecutive Nights); and Difference From Baseline (Adaptation Night)
Description: Sleep Efficiency (SE) is an objective measure of sleep quality derived from polysomnography (PSG); it is a unitless measure defined as the total sleep time (TST) divided by total time in bed (TiB); it can theoretically range from 0 (no sleep at all) to 1 (slept the entire time in bed). Values close to zero indicate very little time spent sleeping while values close to one indicate a large sleep utilization while in bed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: unitless ratio (0 to 1)
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
unitless ratio (0 to 1)
  Baseline SE | 0.72 (0.16) | 0.72 (0.16)
  Sham or Active LFMS (two-night average) | 0.77 (0.11) | 0.79 (0.08)
  Change from Baseline SE | 0.05 (0.11) | 0.07 (0.15)
Statistical Analysis 1: Comparison: Active Low Field Magnetic Stimulation vs Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of SE for active/sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to: H0: Mean changes from Baseline SE for active/sham LFMS are equal Ha: Means differ; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.424, t-test, 2 sided
Statistical Analysis 2: Comparison: Active Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of SE for Baseline and Active LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline SE for Active LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.210, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of SE for Baseline and Sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline SE for Sham LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.190, t-test, 2 sided

5. Primary Outcome: Ease of Sleep (EOS) After Sham vs. Active LFMS (Each Averages of Two Consecutive Nights); and Difference From Baseline (Adaptation Night)
Description: Ease of Sleep (EOS) is assessed after each night as a subjective measure; participants self-rate their ease to fall asleep on a visual analog scale 0-100mm where 0mm is associated with not easy at all (no sleep) and 100mm is associated with no problems to fall asleep. EOS is a proxy measure for a participants sleepiness.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale (0-100mm)
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
units on a scale (0-100mm)
  Baseline EOS | 63.30 (30.99) | 63.30 (30.99)
  Sham or Active LFMS (two-night average) | 51.95 (26.47) | 47.70 (17.76)
  Change from Baseline EOS | -11.35 (25.70) | -15.60 (26.17)
Statistical Analysis 1: Comparison: Active Low Field Magnetic Stimulation vs Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of EOS for active/sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to: H0: Mean changes from Baseline EOS for active/sham LFMS are equal Ha: Means differ; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.535, t-test, 2 sided
Statistical Analysis 2: Comparison: Active Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of EOS for Baseline and Active LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline EOS for Active LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.196, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of EOS for Baseline and Sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline EOS for Sham LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.092, t-test, 2 sided

6. Primary Outcome: MUSC Sleep Quality Score (SQS) After Sham vs. Active LFMS (Each Averages of Two Consecutive Nights); and Difference From Baseline (Adaptation Night)
Description: MUSC Sleep Quality Score (SQS) is assessed after each night as a subjective measure; participants self-rate their perceived sleep quality on a 0-6 scale where 0 is associated with extremely poor sleep quality and 6 is associated with extremely good sleep quality.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (0-6)
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
score on a scale (0-6)
  Baseline SQS | 1.90 (0.74) | 1.90 (0.74)
  Sham or Active LFMS (two-night average) | 2.75 (0.82) | 2.75 (1.25)
  Change from Baseline SQS | 0.85 (0.71) | 0.85 (1.13)
Statistical Analysis 1: Comparison: Active Low Field Magnetic Stimulation vs Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of SQS for active/sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to: H0: Mean changes from Baseline SQS for active/sham LFMS are equal Ha: Means differ; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 1.00, t-test, 2 sided
Statistical Analysis 2: Comparison: Active Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of SQS for Baseline and Active LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline SQS for Active LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.004, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of SQS for Baseline and Sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline SQS for Sham LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.042, t-test, 2 sided

7. Secondary Outcome: Number of Awakenings (#Awake) After Sham vs. Active LFMS (Each Averages of Two Consecutive Nights); and Difference From Baseline (Adaptation Night)
Description: Number of Awakenings (#awake) is the integer number of nocturnal awakenings after initial sleep onset, i.e. a count.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
awakenings
  Baseline #awake | 19 (8.31) | 19 (8.31)
  Sham or Active LFMS (two-night average): number analyzed (Participants) | 10 | 9
  Sham or Active LFMS (two-night average) | 17.45 (5.36) | 21.17 (8.31)
  Change from Baseline #awake: number analyzed (Participants) | 10 | 9
  Change from Baseline #awake | -1.55 (5.30) | 2.50 (6.53)
Statistical Analysis 1: Comparison: Active Low Field Magnetic Stimulation vs Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of #awake for active/sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to: H0: Mean changes from Baseline #awake for active/sham LFMS are equal Ha: Means differ; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Active Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of #awake for Baseline and Active LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline #awake for Active LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.379, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of #awake for Baseline and Sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline #awake for Sham LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.284, t-test, 2 sided

8. Secondary Outcome: Fatigue After Sham vs. Active LFMS (Each Averages of Two Consecutive Nights); and Difference From Baseline (Adaptation Night)
Description: Participants rate after each night how fatigued they feel on a 0-100mm continuous scale; 0mm not at all; 100mm very/a lot.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale (0-100mm)
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
units on a scale (0-100mm)
  Baseline fatigue | 58.10 (24.73) | 58.10 (24.73)
  Sham or Active LFMS (two-night average) | 52.65 (22.30) | 45.45 (27.58)
  Change from Baseline fatigue | -5.45 (11.13) | -12.65 (23.90)
Statistical Analysis 1: Comparison: Active Low Field Magnetic Stimulation vs Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of Fatigue for active/sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to: H0: Mean changes from Baseline Fatigue for active/sham LFMS are equal Ha: Means differ; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.226, t-test, 2 sided
Statistical Analysis 2: Comparison: Active Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of Fatigue for Baseline and Active LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline Fatigue for Active LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.156, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of Fatigue for Baseline and Sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline Fatigue for Sham LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.117, t-test, 2 sided

9. Secondary Outcome: Concentration After Sham vs. Active LFMS (Each Averages of Two Consecutive Nights); and Difference From Baseline (Adaptation Night)
Description: Participants rate after each night their ability to concentrate on a 0-100mm continuous scale; 0mm not at all; 100mm very/a lot. This is a subjective proxy measure for a restorative sleep / sleep quality.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale (0-100mm)
Arm/Group | Active Low Field Magnetic Stimulation | Sham Low Field Magnetic Stimulation
Number analyzed (Participants) | 10 | 10
units on a scale (0-100mm)
  Baseline concentration | 46.80 (22.42) | 46.80 (22.42)
  Sham or Active LFMS (two-night average) | 42.40 (19.58) | 36.80 (20.37)
  Change from Baseline concentration | -4.40 (11.28) | -10.00 (18.09)
Statistical Analysis 1: Comparison: Active Low Field Magnetic Stimulation vs Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of Concentration for active/sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to: H0: Mean changes from Baseline Concentration for active/sham LFMS are equal Ha: Means differ; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.130, t-test, 2 sided
Statistical Analysis 2: Comparison: Active Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of Concentration for Baseline and Active LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline Concentration for Active LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.249, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Low Field Magnetic Stimulation; This is a crossover study; we use a paired t-test to test the hypothesis: H0: Means of Concentration for Baseline and Sham LFMS are equal Ha: Means differ Note this paired t-test is equivalent to a one-sample t-test: H0: Mean changes from Baseline Concentration for Sham LFMS is equal 0 Ha: Mean is not equal zero; Test type: Equivalence — Significance level alpha=0.05; CI=95%; p = 0.114, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Beginning with the baseline adaptation night adverse effect were actively monitored over the duration of the study interventions (distributed over approx. two weeks for each subject); monitoring specifically included all 5 nights spent in the sleep lab (adaptation night #1, first intervention nights 2&3, washout period, and second intervention nights 4&5)
Description: Each study participant was further informed that adverse effects, should they occur outside the active monitoring period and/or after the study concluded, can be reported directly to either the sleep-lab manager, to the attending physician (T. Uhde), or to the clinical psychologist (A. Wilkerson).
Groups:
- Entire Study Population: All participants completed an adaptation night (night #1) in the sleep lab including baseline assessment. Participants were treatment randomized to receive, after the adaptation night in the sleep lab, either two consecutive nights (night #2,#3) of "Active Low Field Magnetic Stimulation" followed by two consecutive nights (night #4,#5) of "Sham Low Field Magnetic Stimulation", or vice versa. A washout period was permitted between nights #3 and #4 when the intervention changed.
  Interventions:
  Active Low Field Magnetic Stimulation A non-invasive form of brain stimulation administered from a device resembling a bird cage. The device covers the top part of the head for the duration of stimulation (20 minutes before sleep)
  Sham Low Field Magnetic Stimulation A simulation of the LFMS-Active intervention, using the same device that produces a sound similar to the sound made by the device during the active treatment, for a similar duration (20 minutes before sleep)
Arm/Group | Entire Study Population
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT03050372/Prot_SAP_000.pdf